CLINICAL TRIAL: NCT03551912
Title: Nigerian Surgical Outcomes Study. A Nigerian, Multi-centre Seven-day Evaluation of Patient Care and Clinical Outcomes for Patients Undergoing Surgery
Brief Title: The Nigerian Surgical Outcomes Study. This Study is Aimed at Observing for Complications Within 30 Days After Surgery
Acronym: NiSOS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Ibadan (Other)
Responsible Party: Principal Investigator, Babatunde Osinaike, Reader, University of Ibadan
Other Study IDs: NHREC/01/01/2007
Record Dates: First submitted 2018-05-26; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery — All patients coming for elective surgery

SUMMARY:
The Nigerian Surgical Outcome Study is a national 30-day observational cohort study of complications after surgery. Various institutions across Nigeria will be involved. The study aims at providing detailed data describing post-operative complications, requirement for intensive care and mortality. All patients undergoing either elective surgery during a 7-day study period with a planned overnight stay will be recruited.

DETAILED DESCRIPTION:
It is widely known that complications after surgery are responsible for a good number of morbidity and mortality following surgery. This national cohort study will help contribute to, and allow a better computation of data on post-operative complications and mortality following elective surgery in Nigeria.

This study therefore has important public health implications for Nigeria. This study will also provide a baseline for other similar studies in future being the first of such in Nigeria.

Objectives are:

1. To determine the mortality rate on the day of surgery for patients undergoing surgery in Nigeria.
2. To determine the in-hospital mortality rate for patients undergoing surgery in Nigeria.
3. To describe the relationship between anaesthetic complications and postoperative mortality.
4. To describe the relationship between postoperative complications and postoperative mortality.
5. To describe the proportional contribution of communicable, non-communicable diseases and traumatic injuries to critical care admissions and in-hospital mortality in Nigeria. We plan to recruit a minimum of 5 centres per state, made up of federal, state and private hospitals. The national coordinating centre shall be the University College Hospital, Ibadan. Regional coordinating centres shall be in Lagos, Kwara, Enugu, Kaduna, Port-Harcourt, Maiduguri and Abuja.The plan is to recruit all eligible patients during the recruitment week.

All recruited patients would have had the routine preoperative surgical and anaesthetic review. Since the study is purely observational, all basic intraoperative procedures as it relates to surgery and anaesthesia will not be altered. Following informed written consent by the patient, the following information will be obtained.

* Results of preoperative Haemoglobin, Total white cell count, and Creatinine.
* Patient's socio-demographics.
* Co-morbid conditions
* Type of anaesthesia and surgical procedure.
* Anaesthetic and Surgical details
* Critical care admission post-operatively, and
* Postoperative complications observed till discharge or up to 30 days if on admission.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients admitted to participating centres undergoing elective surgery with a planned overnight hospital stay following surgery during a seven-day study period. The recruitment week will run between June and July 2018.

Exclusion Criteria:

Patients undergoing planned day-case surgery or procedures outside the operating theatre.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults or Paediatrics coming for elective surgical procedures
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-06-14 (Estimated); Study Completion 2018-08-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative complications | At discharge or 30 days, whichever is earlier.
  In-hospital post-operative complications of any cause

SECONDARY OUTCOMES:
Mortality | Within 24 hours
  Rate of mortality on the day of surgery
Mortality | At 30 days after surgery
  In-hospital all-cause mortality
Critical care admission | At 30 days after surgery
  Critical care admission after surgery
Duration of hospital stay | At discharge or 30 days
  Duration of hospital stay after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Babatunde Babatunde, MBChB,FMCA, Principal Investigator — University of Ibadan/University College Hospital
Locations (1):
- University College Hospital, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: No
Data will be pseudo-anonymised by generation of a unique numeric code and transcribed by local investigators onto an internet based electronic CRF. Each patient will only be identified on the electronic CRF by their numeric code; thus the co- ordinating study team cannot trace data back to an individual patient without contact with the local team.

REFERENCES:
- [Result] Biccard BM, Madiba TE, Kluyts HL, Munlemvo DM, Madzimbamuto FD, Basenero A, Gordon CS, Youssouf C, Rakotoarison SR, Gobin V, Samateh AL, Sani CM, Omigbodun AO, Amanor-Boadu SD, Tumukunde JT, Esterhuizen TM, Manach YL, Forget P, Elkhogia AM, Mehyaoui RM, Zoumeno E, Ndayisaba G, Ndasi H, Ndonga AKN, Ngumi ZWW, Patel UP, Ashebir DZ, Antwi-Kusi AAK, Mbwele B, Sama HD, Elfiky M, Fawzy MA, Pearse RM; African Surgical Outcomes Study (ASOS) investigators. Perioperative patient outcomes in the African Surgical Outcomes Study: a 7-day prospective observational cohort study. Lancet. 2018 Apr 21;391(10130):1589-1598. doi: 10.1016/S0140-6736(18)30001-1. Epub 2018 Jan 3. PMID 29306587
- [Result] International Surgical Outcomes Study group. Global patient outcomes after elective surgery: prospective cohort study in 27 low-, middle- and high-income countries. Br J Anaesth. 2016 Oct 31;117(5):601-609. doi: 10.1093/bja/aew316. PMID 27799174